CLINICAL TRIAL: NCT03126916
Title: A Phase 3 Study of 131I-Metaiodobenzylguanidine (131I-MIBG) or ALK Inhibitor Therapy Added to Intensive Therapy for Children With Newly Diagnosed High-Risk Neuroblastoma (NBL)
Brief Title: Testing the Addition of 131I-MIBG or Lorlatinib to Intensive Therapy in People With High-Risk Neuroblastoma (NBL)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANBL1531; NCI-2016-01734 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANBL1531 (Other: Children's Oncology Group); ANBL1531 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Ganglioneuroblastoma; Ganglioneuroblastoma, Nodular; Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma; Neuroblastoma | interventions — Stem Cell Transplantation; Specimen Handling; Biopsy; Busulfan; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Dexrazoxane; Razoxane; dinutuximab; Doxorubicin; etoposide phosphate; Congresses as Topic; Radiation; 3-Iodobenzylguanidine; Isotretinoin; lorlatinib; Magnetic Resonance Spectroscopy; Melphalan; sargramostim; Colony-Stimulating Factors; Thiotepa; Topotecan; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (chemotherapy, HSCT, EBRT) (Experimental): See Arm A in detailed description.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Dexrazoxane Hydrochloride; Biological: Dinutuximab; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Drug: Etoposide Phosphate; Radiation: External Beam Radiation Therapy; Radiation: Iobenguane I-123; Drug: Isotretinoin; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Biological: Sargramostim; Procedure: Therapeutic Conventional Surgery; Drug: Thiotepa; Drug: Topotecan Hydrochloride; Drug: Vincristine Sulfate
- Arm B (Iobenguane I-131, chemotherapy, HSCT, EBRT) (Experimental): See Arm B in detailed description.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Dexrazoxane Hydrochloride; Biological: Dinutuximab; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Drug: Etoposide Phosphate; Radiation: External Beam Radiation Therapy; Radiation: Iobenguane I-123; Radiation: Iobenguane I-131; Drug: Isotretinoin; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Biological: Sargramostim; Procedure: Therapeutic Conventional Surgery; Drug: Thiotepa; Drug: Topotecan Hydrochloride; Drug: Vincristine Sulfate
- Arm C (Iobenguane I-131, chemotherapy, BuMel, HSCT, EBRT) (Experimental): See Arm C in detailed description. Closed to accrual as of 12/17/20.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Busulfan; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Dexrazoxane Hydrochloride; Biological: Dinutuximab; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Drug: Etoposide Phosphate; Radiation: External Beam Radiation Therapy; Radiation: Iobenguane I-131; Drug: Isotretinoin; Procedure: Magnetic Resonance Imaging; Drug: Melphalan Hydrochloride; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Biological: Sargramostim; Procedure: Therapeutic Conventional Surgery; Drug: Thiotepa; Drug: Topotecan Hydrochloride; Drug: Vincristine Sulfate
- Arm D (chemotherapy, HSCT, EBRT) (Experimental): See Arm D in detailed description.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Dexrazoxane Hydrochloride; Biological: Dinutuximab; Drug: Doxorubicin Hydrochloride; Drug: Etoposide Phosphate; Radiation: External Beam Radiation Therapy; Radiation: Iobenguane I-123; Drug: Isotretinoin; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Biological: Sargramostim; Procedure: Therapeutic Conventional Surgery; Drug: Thiotepa; Drug: Topotecan Hydrochloride; Drug: Vincristine Sulfate
- Arm E (lorlatinib, chemotherapy, HSCT, EBRT) (Experimental): See Arm E in detailed description.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Dexrazoxane Hydrochloride; Biological: Dinutuximab; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Drug: Etoposide Phosphate; Radiation: External Beam Radiation Therapy; Radiation: Iobenguane I-123; Drug: Isotretinoin; Drug: Lorlatinib; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Biological: Sargramostim; Procedure: Therapeutic Conventional Surgery; Drug: Thiotepa; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous HSCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Busilvex; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
  Arms: Arm C (Iobenguane I-131, chemotherapy, BuMel, HSCT, EBRT)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm A (chemotherapy, HSCT, EBRT); Arm B (Iobenguane I-131, chemotherapy, HSCT, EBRT); Arm D (chemotherapy, HSCT, EBRT); Arm E (lorlatinib, chemotherapy, HSCT, EBRT)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Dexrazoxane Hydrochloride — Given IV
  Other Names: Cardioxane; Totect; Zinecard
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; Dinutuximab Beta; MOAB Ch14.18; monoclonal antibody Ch14.18; Qarziba; Unituxin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
  Arms: Arm A (chemotherapy, HSCT, EBRT); Arm B (Iobenguane I-131, chemotherapy, HSCT, EBRT); Arm C (Iobenguane I-131, chemotherapy, BuMel, HSCT, EBRT); Arm E (lorlatinib, chemotherapy, HSCT, EBRT)
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Radiation: Iobenguane I-123 — Given 123 I-MIBG
  Other Names: 123I-Metaiodobenzylguanidine; 123I-MIBG; AdreView; I-123-MIBG; Iobenguane (123 I); Iobenguane I 123; Iodine I 123-Metaiodobenzylguanidine; MIBG I-123
  Arms: Arm A (chemotherapy, HSCT, EBRT); Arm B (Iobenguane I-131, chemotherapy, HSCT, EBRT); Arm D (chemotherapy, HSCT, EBRT); Arm E (lorlatinib, chemotherapy, HSCT, EBRT)
Radiation: Iobenguane I-131 — Given IV
  Other Names: (131)I-MIBG; 131I-MIBG; I 131 Meta-iodobenzylguanidine; I-131 Metaiodobenzylguanidine; Iobenguane (131I); Iobenguane I 131; Iodine I 131 Metaiodobenzylguanidine; MIBG I-131; Raiatt MIBG-I 131
  Arms: Arm B (Iobenguane I-131, chemotherapy, HSCT, EBRT); Arm C (Iobenguane I-131, chemotherapy, BuMel, HSCT, EBRT)
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Absorica; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Myorisan; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret; ZENATANE
Drug: Lorlatinib — Given PO
  Other Names: 2H-4,8-Methenopyrazolo(4,3-H)(2,5,11)benzoxadiazacyclotetradecine-3-carbonitrile, 7-amino-12-fluoro-10,15,16,17-tetrahydro-2,10,16-trimethyl-15-oxo-, (10R)-; Lorbrena; Lorviqua; PF 06463922; PF-06463922; PF06463922
  Arms: Arm E (lorlatinib, chemotherapy, HSCT, EBRT)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Arm B (Iobenguane I-131, chemotherapy, HSCT, EBRT); Arm C (Iobenguane I-131, chemotherapy, BuMel, HSCT, EBRT); Arm D (chemotherapy, HSCT, EBRT)
Drug: Melphalan Hydrochloride — Given IV
  Other Names: Alkeran; Alkerana; Evomela; Hepzato
  Arms: Arm C (Iobenguane I-131, chemotherapy, BuMel, HSCT, EBRT)
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgery
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; SH 105; SH-105; SH105; STEPA; Tepadina; Tepylute; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Evotopin; Hycamptamine; Hycamtin; Nogitecan Hydrochloride; Potactasol; SKF S 104864 A; SKF S-104864-A; SKF S104864A; Topotec; Topotecan HCl; topotecan hydrochloride (oral)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Arm A (chemotherapy, HSCT, EBRT); Arm B (Iobenguane I-131, chemotherapy, HSCT, EBRT); Arm C (Iobenguane I-131, chemotherapy, BuMel, HSCT, EBRT); Arm D (chemotherapy, HSCT, EBRT)

SUMMARY:
This phase III trial studies iobenguane I-131 or lorlatinib and standard therapy in treating younger patients with newly-diagnosed high-risk neuroblastoma or ganglioneuroblastoma. Radioactive drugs, such as iobenguane I-131, may carry radiation directly to tumor cells and not harm normal cells. Lorlatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving iobenguane I-131 or lorlatinib and standard therapy may work better compared to lorlatinib and standard therapy alone in treating younger patients with neuroblastoma or ganglioneuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine in the context of a randomized trial whether the event-free survival (EFS) of patients with newly diagnosed high-risk neuroblastoma (NBL) is improved with the addition of iobenguane I-131 (131I-MIBG) during induction, prior to tandem autologous stem cell transplantation (ASCT).

II. To determine whether the addition of lorlatinib to intensive multimodality therapy for patients with high-risk NBL whose tumors harbor activating point mutations in the ALK gene with a variant allele frequency (VAF) >= 5% results in superior EFS compared to a contemporaneously treated cohort of patients with tumors without documented ALK activating mutations.

SECONDARY OBJECTIVES:

I. To describe the toxicities associated with treatment for high-risk NBL with and without the addition of 131I-MIBG or ALK inhibitor therapy.

II. To estimate EFS and describe toxicity in patients with newly diagnosed high-risk NBL randomized to treatment with an 131I-MIBG-containing induction prior to busulfan/melphalan (BuMel) ASCT.

III. To describe the overall survival (OS) and response rates (evaluated per International Neuroblastoma Response Criteria [INRC] criteria prior to ASCT and prior to post-consolidation therapy) for patients with high-risk neuroblastoma treated with or without 131I-MIBG or ALK inhibitor therapy.

IV. To prospectively evaluate the relationship of response rate per revised International Neuroblastoma Response Criteria (INRC) to EFS and OS in patients with high-risk NBL treated with and without the addition of 131I-MIBG or ALK inhibitor therapy.

EXPLORATORY OBJECTIVES:

I. To evaluate whole body radiation dose, tumor factors, and host factors as potential predictors of efficacy and/or toxicity associated with 131I-MIBG therapy and transplant conditioning.

II. To describe end-Induction response, EFS, and OS according to specific ALK mutations, VAF, ALK amplification, the presence of additional genomic findings, or the ALK inhibitor administered.

III. To characterize changes in tumor markers (circulating tumor deoxyribonucleic acid [DNA], including ALK and other tumor specific genetic aberrations, and circulating GD2) over time in response to protocol therapy.

IV. To correlate results of tumor and host profiling with end-induction response and EFS.

V. To prospectively evaluate EFS for patients with MIBG non-avid high-risk NBL compared to patients with MIBG-avid high-risk NBL who are randomized to treatment without 131I-MIBG.

VI. To correlate Curie scores calculated from 131I-MIBG post-treatment scans with end-induction response, EFS and OS.

VII. To describe changes in image defined risk factors (IDRFs) over the course of induction therapy, with correlation to surgical outcomes and local failure rates following primary tumor resection.

VIII. To define patterns of failure at time of first relapse or progression in patients with high-risk NBL.

IX. To determine the feasibility of prospectively monitoring adverse events using electronic health records.

X. To compare local, central, and computer assisted Curie score assignment at baseline and during therapy in patients with MIBG-avid high-risk NBL.

XI. To compare late toxicities (including impaired organ function and secondary tumor occurrence) in patients treated with 131I-MIBG or ALK inhibitor therapy to late toxicities in patients who have not received these therapies.

XII. To determine the association between household material hardship (HMH) and clinical outcomes, including event free and overall survival, and 131I-MIBG receipt.

XIII. To compare the outcomes (EFS, OS, and toxicity) of patients treated with post-consolidation therapy that does not contain aldesleukin to historical outcome data for patients treated with similar induction and consolidation regimens followed by post-consolidation therapy that contained aldesleukin.

XIV. To characterize and describe longitudinal neuropsychological and behavioral effects of high-risk neuroblastoma therapy.

XV. To evaluate change in neurobehavioral outcomes over time in patients with neuroblastoma treated with high-risk neuroblastoma therapy plus lorlatinib compared to high-risk therapy alone using parent- or self-report measures of adaptive, executive, and psychosocial functioning.

XVI. To characterize the pharmacokinetics and pharmaceutical properties of lorlatinib in children with high-risk neuroblastoma.

XVII. To compare the EFS of patients enrolled on Arm E and treated with lorlatinib to the EFS of a historical control comprised of patients with ALK aberrant disease treated on ANBL0532 (NCT00567567).

XVIII. To describe the EFS of patients enrolled on Arm E according to lorlatinib exposure during post-consolidation.

OUTLINE: Patients are randomized or assigned to 1 of 5 arms.

All patients receive cyclophosphamide intravenously (IV) over 15-30 minutes and topotecan hydrochloride IV over 30 minutes on days 1-5 during cycle 1 of induction therapy in the absence of disease progression or unacceptable toxicity. Patients not assigned to an Arm by the end of cycle 1 may receive an addition cycle of cyclophosphamide and topotecan.

ARM A (CLOSED TO ACCRUAL AS OF SEPTEMBER 28, 2023):

INDUCTION THERAPY: Patients receive cyclophosphamide IV over 15-30 minutes and topotecan hydrochloride IV over 30 minutes on days 1-5 of cycle 2 and cisplatin IV over 4 hours and etoposide phosphate IV over 2 hours on days 1-3 of cycles 3 and 5. Patients also receive vincristine sulfate IV over 1 minute on day 1 and dexrazoxane hydrochloride IV over 5-15 minutes, doxorubicin hydrochloride IV over 1-15 minutes, and cyclophosphamide IV over 1-6 hours on days 1-2 of cycle 4 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION THERAPY:

HSCT#1: Patients receive thiotepa IV over 2 hours on days -7 to -5 and cyclophosphamide IV over 1 hour on days -5 to -2 in the absence of disease progression or unacceptable toxicity.

HSCT#2: Patients receive melphalan hydrochloride IV over 30 minutes on days -7 to -5, and etoposide phosphate IV over 24 hours and carboplatin IV over 24 hours on days -7 to -4 in the absence of disease progression or unacceptable toxicity.

POST-CONSOLIDATION THERAPY: Patients receive sargramostim subcutaneously (SC) on days 1-14, dinutuximab IV over 10 hours on days 4-7 of cycles 1-5, and isotretinoin orally (PO) twice daily (BID) on days 11-24 of cycles 1-5, and days 15-28 during cycle 6 in the absence of disease progression or unacceptable toxicity.

Patients undergo echocardiography or multigated acquisition (MUGA) scan, magnetic resonance imaging (MRI) or computed tomography (CT) scan, receive 123I-MIBG and undergo MIBG imaging, bone marrow aspiration and biopsy and blood sample collection throughout the study.

ARM B (CLOSED TO ACCRUAL AS OF SEPTEMBER 28, 2023):

INDUCTION THERAPY: Patients receive cyclophosphamide, topotecan hydrochloride, cisplatin, and etoposide phosphate as in Arm A, iobenguane I-131 IV over 1.5-2 hours on day 1 beginning 3 weeks after the start of cycle 3, and vincristine sulfate, dexrazoxane hydrochloride, doxorubicin hydrochloride, and cyclophosphamide as in Arm A beginning no sooner than 35 days after the infusion of iobenguane I-131.

CONSOLIDATION THERAPY:

HSCT#1: Patients receive thiotepa and cyclophosphamide as in Arm A.

HSCT#2: Patients receive melphalan, etoposide phosphate, and carboplatin as in Arm A.

POST-CONSOLIDATION THERAPY: Patients receive sargramostim, dinutuximab, and isotretinoin as in Arm A-D.

Patients undergo echocardiography or MUGA scan, MRI or CT scan, receive 123I-MIGB and undergo MIBG imaging, bone marrow aspiration and biopsy and blood sample collection throughout the study.

ARM C (CLOSED TO ACCRUAL AS OF DECEMBER 17, 2020):

INDUCTION THERAPY: Patients receive cyclophosphamide, topotecan hydrochloride, cisplatin, etoposide phosphate, iobenguane I-131, vincristine sulfate, dexrazoxane hydrochloride, doxorubicin hydrochloride, and cyclophosphamide as in Arm B.

CONSOLIDATION THERAPY: Patients receive busulfan IV over 3 hours on days -6 to -3 and melphalan hydrochloride IV over 30 minutes on day -1 in the absence of disease progression or unacceptable toxicity.

POST-CONSOLIDATION THERAPY: Patients receive sargramostim, dinutuximab, and isotretinoin as in Arm A.

Patients undergo echocardiography or MUGA scan, MRI or CT scan, receive 123I-MIGB and undergo MIBG imaging, bone marrow aspiration and biopsy and blood sample collection throughout the study.

ARM D (CLOSED TO ACCRUAL AS OF SEPTEMBER 28, 2023): Patients receive treatment identical to Arm A.

Patients undergo echocardiography or MUGA scan, MRI or CT scan, receive 123I-MIGB and undergo MIBG imaging, bone marrow aspiration and biopsy and blood sample collection throughout the study and may undergo fludeoxyglucose- positron emission tomography (PET) scan on study.

ARM E:

INDUCTION THERAPY: Patients receive cyclophosphamide, topotecan hydrochloride, cisplatin, etoposide phosphate, vincristine sulfate, dexrazoxane hydrochloride, doxorubicin hydrochloride, and cyclophosphamide as in Arm A. Patients also receive lorlatinib PO once daily (QD) starting with cycle 2 and continue until HSCT #1 in the absence of disease progression or unacceptable toxicity. For patients transferring from ANBL2131 (NCT06172296) to ANBL1531 (NCT03126916) Arm E, protocol therapy on ANBL1531 (NCT03126916) begins with induction cycle 2 on Arm E (topotecan, cyclophosphamide and lorlatinib).

CONSOLIDATION THERAPY:

HSCT#1: Patients receive thiotepa and cyclophosphamide as in Arm A. Patients also receive lorlatinib PO QD until day -8 of HSCT#2 in the absence of disease progression or unacceptable toxicity.

HSCT#2: Patients receive melphalan hydrochloride, etoposide phosphate, carboplatin as in Arm A. Lorlatinib is restarted when patient has reached at least day +14 post-HSCT#2 and is able to tolerate enteral medications, provided there is no evidence of disease progression or unacceptable toxicity.

RADIATION THERAPY: Patients receive lorlatinib PO QD concurrently with radiation therapy in the absence of disease progression or unacceptable toxicity.

POST-CONSOLIDATION THERAPY: Patients receive sargramostim and dinutuximab as in Arm A-D. Patients also receive isotretinoin PO BID on days 11-24 of cycles 1-5 and days 15-28 of cycle 6, and lorlatinib PO QD on days 15-28 of cycles 2-5 and days 1-28 of cycle 6 in the absence of disease progression or unacceptable toxicity.

CONTINUATION THERAPY: Patients receive lorlatinib PO QD on days 1-28. Cycles repeat every 28 days for 18 months in the absence of disease progression or unacceptable toxicity.

Patients undergo echocardiography or MUGA scan, MRI or CT scan, undergo MIBG imaging, bone marrow aspiration and biopsy and blood sample collection throughout the study and may undergo PET scan on study.

After completion of study therapy, patients in Arms A-D are followed up every 3 months for 18 months, and then every 6 months for 42 months; patients in Arm E are followed up every 3 months for 6 months, and then every 6 months for 42 months.

ELIGIBILITY:
Inclusion Criteria:

* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Patients must be enrolled on ANBL00B1 (NCT00904241) or APEC14B1 (NCT02402244) prior to enrollment on ANBL1531 (NCT03126916)
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Patient must be >= 365 days and =< 30 years of age at diagnosis
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Patients must have a diagnosis of neuroblastoma or ganglioneuroblastoma (nodular) verified by tumor pathology analysis or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites; the following disease groups are eligible:

  * Patients with International Neuroblastoma Risk Group (INRG) stage M disease are eligible if found to have either of the following features:

    * MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of additional biologic features; OR
    * Age > 547 days regardless of biologic features
  * Patients with INRG stage MS disease with MYCN amplification
  * Patients with INRG stage L2 disease with MYCN amplification
  * Patients > 547 days of age initially diagnosed with INRG stage L1, L2 or MS disease who progressed to stage M without prior chemotherapy may enroll within 4 weeks of progression to stage M
  * Patients >= 365 days of age initially diagnosed with MYCN amplified INRG stage L1 disease who progress to stage M without systemic therapy may enroll within 4 weeks of progression to stage M
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Patients initially recognized to have high-risk disease must have had no prior systemic therapy (other than topotecan/cyclophosphamide initiated on an emergent basis and within allowed timing); patients observed or treated with a single cycle of chemotherapy per a low or intermediate risk neuroblastoma regimen (e.g., as per ANBL0531, ANBL1232 or similar) for what initially appeared to be non-high risk disease but subsequently found to meet the criteria will also be eligible; patients who receive localized emergency radiation to sites of life-threatening or function-threatening disease prior to or immediately after establishment of the definitive diagnosis will be eligible
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/sex as follows:

  * 1 to < 2 years: male = 0.6; female = 0.6
  * 2 to < 6 years: male = 0.8; female = 0.8
  * 6 to < 10 years: male = 1; female = 1
  * 10 to < 13 years: male = 1.2; female = 1.2
  * 13 to < 16 years: male = 1.5; female = 1.4
  * >= 16 years: male = 1.7; female = 1.4
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Total bilirubin =< 1.5 x upper limit of normal (ULN) for age, and
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 10 x ULN; for the purposes of this study, ULN for SGPT (ALT) is 45
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Shortening fraction of >= 27% by echocardiogram, or ejection fraction of > 50% by echocardiogram or radionuclide angiogram
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: No known contraindication to peripheral blood stem cell (PBSC) collection; examples of contraindications might be a weight or size less than the collecting institution finds feasible, or a physical condition that would limit the ability of the child to undergo apheresis catheter placement (if necessary) and/or the apheresis procedure
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): See ANBL2131 (NCT06172296) protocol for eligible high-risk neuroblastoma diagnoses
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): In addition, all patients transferring from ANBL2131 (NCT06172296) to ANBL1531 (NCT03126916) Arm E must have tumors with an ALK aberration
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Given the lack of data with lorlatinib in infant populations, patients transferring from ANBL2131 (NCT06172296) to ANBL1531 (NCT03126916) must be > 1 year of age at time of transfer to ANBL1531 (NCT03126916). Patients < 1 year of age found to have a qualifying ALK alteration as part of ANBL2131 (NCT06172296) may continue to participate in ANBL2131 (NCT06172296)
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Patients initially recognized to have high-risk disease must have received no more than one cycle of topotecan/cyclophosphamide either after enrollment to ANBL2131 (NCT06172296) or started emergently prior to enrollment to ANBL2131 (NCT06172296)
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Patients may have received up to one cycle of intermediate risk chemotherapy prior to initial enrollment to ANBL2131 (NCT06172296)
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Patients may have received localized emergency radiation to sites of life-threatening or function-threatening disease prior to or immediately after establishment of the definitive diagnosis
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): In order to facilitate patient transfer and ensure timely distribution of lorlatinib, there are no blood count requirements to meet at time of transfer from ANBL2131 (NCT06172296) to ANBL1531 ((NCT03126916) Arm E. Note the blood count criteria that must be met prior to start of Induction cycle 2 on Arm E. Lorlatinib therapy should start no sooner than day 1 of Induction cycle 2
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): No known irreversible grade 2 or greater atrioventricular (AV) block
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Due the potential psychiatric risks from lorlatinib, patients should not have a personal history of a serious psychiatric disorder requiring pharmacologic intervention or severe enough to be considered life-threatening
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): No known contraindication to PBSC collection. Examples of contraindications might be a weight or size less than the collecting institution deems feasible, or a physical condition that would limit the ability of the child to undergo apheresis catheter placement (if necessary) and/or the apheresis procedure

Exclusion Criteria:

* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Patients with INRG stage L2 tumors without amplification of MYCN regardless of tumor histology (may meet criteria for high risk classification but are not eligible for this trial)
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Patients with bone marrow failure syndromes
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Patients for whom targeted radiopharmaceutical therapy would be contraindicated due to underlying medical disorders
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs; a pregnancy test is required for female patients of childbearing potential
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Lactating females who plan to breastfeed their infants
* FOR PATIENTS ENROLLING TO ANBL1531 (NCT03126916) WITHOUT PRIOR ANBL2131 (NCT06172296) ENROLLMENT: Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Patients who have previously received treatment with lorlatinib or other ALK inhibitor
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Patients who have undergone treatment arm randomization callback or started induction cycle 2 on ANBL2131 (NCT06172296)
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Patients who have an INRG Stage L2 tumor without amplification of MYCN regardless of tumor histology (may meet criteria for high risk classification but are not eligible for this trial)
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Patients with bone marrow failure syndromes
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Lactating females who plan to breastfeed their infants
* PATIENTS WITH TUMORS HARBORING ALK ALTERATIONS TRANSFERRING TO ANBL1531 (NCT03126916) ARM E FROM ANBL2131 (NCT06172296) (EFFECTIVE WITH AMENDMENT 13C): Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation

Ages: 365 Days to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 750 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) (Arm A, B, D, and E) | 3 years
  EFS time is calculated from date of randomization or assignment to first episode of disease relapse or progression, second malignancy, or death, or until last contact if no event has occurred.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 18 months for Arms A-D and 28 months for Arm E
  The proportion of patients with at least one Grade 3 or higher toxicity during protocol therapy, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, will be reported.
EFS (Arm C) | 3 years
  EFS time is calculated from date of randomization to first episode of disease relapse or progression, second malignancy, or death, or until last contact if no event has occurred.
Overall survival (OS) | 3 years
  OS time is calculated from date of randomization or assignment until death, or until last contact if patient is alive.
Response rate | Up to 6 months
  The response rate will be calculated among all evaluable patients at end-Induction. Responders are defined as patients who achieve a >= partial response (PR) per the revised International Neuroblastoma Response Criteria (INRC).

CONTACTS AND LOCATIONS:
Overall Officials: Steven G DuBois, Principal Investigator — Children's Oncology Group
Locations (161):
- United States (151):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (9):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico

REFERENCES:
- [Derived] Weiss BD, Yanik G, Naranjo A, Zhang FF, Fitzgerald W, Shulkin BL, Parisi MT, Russell H, Grupp S, Pater L, Mattei P, Mosse Y, Lai HA, Jarzembowski JA, Shimada H, Villablanca JG, Giller R, Bagatell R, Park JR, Matthay KK. A safety and feasibility trial of 131 I-MIBG in newly diagnosed high-risk neuroblastoma: A Children's Oncology Group study. Pediatr Blood Cancer. 2021 Oct;68(10):e29117. doi: 10.1002/pbc.29117. Epub 2021 May 24. PMID 34028986